CLINICAL TRIAL: NCT02977988
Title: Neural Mechanisms in Women's Treatment and Early Recovery
Brief Title: Women's Treatment and Early Recovery
Acronym: MBRP-W
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, David S Black, PhD, Associate Professor of Public Health Sciences, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UP-14-00391-AM001; 5R01DA038648-04 (NIH)
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Substance-related Disorders
Keywords: Mindfulness; Women; Relapse prevention; Clinical trial; Substance use disorder; Ethnically diverse; Underserved; Health disparities; Stress; Addiction; Latina/Hispanic; African American; Treatment retention; Residential treatment; Brain Imaging
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive | interventions — Mindfulness; Salvage Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Meditation (Experimental): Mindfulness-Based Relapse Prevention-Women (MBRP-W)
  Interventions: Behavioral: Mindfulness Meditation
- Active Comparator (Active Comparator): Brain and Recovery (B&R)
  Interventions: Behavioral: Brain and Recovery (B&R)

INTERVENTIONS:
Behavioral: Mindfulness Meditation — MBRP-W is delivered in 12 bi-weekly 80-minute group sessions. Facilitators with previous experience in MBSR and trained in MBRP-W will deliver each group. Each session has a central theme and is divided into five segments consisting of: (a) a welcome meditation or other mindfulness practice, (b) a review of session objectives, (c) a brief didactic psycho-educational presentation and discussion based on the session's theme, (d) experiential and formal meditation or other practices, and (e) readings and assignments for the next class. Participants are expected to learn skill building techniques to reducing stress using mindfulness-based principles to complement their recovery treatment program.
  Other Names: Mindfulness-Based Relapse Prevention-Women (MBRP-W)
  Arms: Mindfulness Meditation
Behavioral: Brain and Recovery (B&R) — B&R is delivered in 12 bi-weekly 80-minute group sessions delivered by two trained interventionists. The B&R group will receive didactic education on the neurobiology of addiction. B&R contains no information on behavior change, stress reduction, or mindfulness-based or relapse-related content. The intervention was developed over three years with a population similar to those in the study and with input from patients and experts on neurobiology of addiction. Topics include: (1) brain structures and functions related to addiction, (2) effects of various types of substances on the brain, and (3) rewarding effects and how these lead to addiction. Participants are expected to gain knowledge pertaining to the effects of drugs on the brain.
  Arms: Active Comparator

SUMMARY:
Approximately 25 million Americans struggle with alcohol or drug problems annually. Abuse of alcohol and drugs is costly to our nation, exacting more than $428 billion in costs related to crime, lost work productivity and health care. While effective treatments exist, over half of those who enter treatment for substance use disorders drop out early in treatment and return to alcohol or drug abuse. Psychological stress is a causal factor in the pathogenesis of substance use disorder (SUD) and relapse risk. Low-income women report high levels of stress in SUD residential treatment stemming from significant economic and family stressors in addition to challenges of adjusting to residential treatment demands. Unmanaged stress, especially in early stages of residential treatment, is a major concern because it can increase dropout. Dropout from residential treatment places women at risk of substance use relapse. A gap in knowledge persists regarding the use of mindfulness-based interventions with racially/ethnically diverse low-income women with SUDs, especially regarding the efficacy of adapted (Mindfulness-based interventions) MBIs for preventing residential dropout and decreasing relapse. We have fully adapted, developed, and pilot tested a novel MBI, Moment-by-Moment in Women's Recovery: Mindfulness Based Relapse Prevention for Women (MBRP-W), that supports the needs of women in residential treatment. This MBI integrates relapse prevention, addresses literacy level, and is relevant to issues surrounding treatment- and relapse-related stressors of disadvantaged women. The current project has three specific aims: (1) to test the efficacy of MBRP-W on residential treatment retention and substance use relapse in racially/ethnically diverse low-income women; (2) to determine the mechanisms of change underlying the MBRP-W program; and (3) to explore neural changes associated with program effects. A rationale for MBRP-W is the need for self-initiated stress management skills in women with SUDs during the early stressful periods of residential treatment that increase risk of dropout and relapse.

DETAILED DESCRIPTION:
* This randomized clinical trial will deliver two interventions as add-ons to residential substance use disorder (SUD) treatment: (1) Moment-by-Moment in women's Recovery: Mindfulness-Based Approach to Relapse Prevention (MBRP-W) and (2) Brain and Recovery (B&R) which serves as an active psychoeducational attention control group.
* Participants (N=165) who meet study eligibility criteria based on intake assessment will be recruited and complete baseline assessments during weeks 3-6 after entry into a residential treatment program. Participants will be randomly assigned to interventions using Urn randomization. All participants (MBRP-W and B&R) will receive SUD treatment as normally provided by the treatment program. Fifteen participants from each intervention group (N=30) will be selected to participate in a brain imaging (MRI and fMRI) substudy.
* Participants will be adult females who have been admitted to a residential treatment center in an urban area of California and who are diagnosed with a SUD based on clinical intake Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V) diagnostic assessment.
* MBRP-W is delivered in 12 bi-weekly 80-minute group sessions with SUD clinical populations. Facilitators will have previous experience in MBSR facilitation and will be trained in MBRP-W. Each session has a central theme and is divided into five segments consisting of (a) a welcome meditation or other mindfulness practice, (b) a review of session objectives, (c) a brief didactic psycho-educational presentation and discussion based on the session's theme, (d) experiential and formal meditation or other practices, and (e) readings and practice assignments for the next class.
* B&R is delivered in 12 bi-weekly 80-minute group sessions with SUD clinical populations. Facilitators will be trained in B&R. The B&R group will receive didactic education on the neurobiology of addiction. B&R contains no information on behavior change, relapse prevention, stress reduction, or mindfulness-based or relapse-related content. The intervention was developed over three years with a population similar to that of the current study (i.e., racially/ethnically diverse and low-income women in SUD treatment) with input and review from focus group participants, care providers in SUD treatment, and three experts on the neurobiology of addiction. Topics include: (1) brain structure and function related to addiction, (2) effects of various types of substance use on the brain, and (3) rewarding effects of substance use and how these rewarding effects can lead to addiction.
* There are three data collection points, 1) baseline, 2) immediate post-intervention, and 3) 8-months post-intervention completion. Data will be collected in-person by research interviewers via computer-assisted interviews, which includes administration of an alcohol Breathalyzer test to assess alcohol use and collection of a urine sample to assess drug use. Interviews will be conducted at the treatment program (for those who remain in residential treatment) or at convenient locations for participants no longer in treatment. Baseline interview will occur prior to randomization, post-intervention interview will occur within 1-2 weeks of the last group session, and the follow-up interview will occur at an 8-months post-intervention completion window. Brain imaging for a subsample of participants will be completed at baseline and immediate post-intervention.
* Number of intervention program class sessions attended will be collected for all enrolled participants.
* Participant Satisfaction Surveys measuring acceptability, credibility, and perceived utility of the study arms will be administered to both groups at two class sessions.
* Applied Mindfulness Practice Scale (AMPS) measuring the participant's application of mindfulness skills to address life challenges, will be administered to the MBRP-W participants at four class sessions as well as at follow-up. Mindfulness practice effort will also be assessed at these same four class sessions.
* An in-treatment clinical record review of services will be collected weekly for the duration of residential treatment.

ELIGIBILITY:
Inclusion criteria for parent study:

* Female
* Adult in California (18 years or older)
* Diagnosed with a substance use disorder (SUD)
* Speaks fluent English
* Client at study site, substance use disorder residential facility at time of recruitment

Exclusion criteria for parent study:

* Inability to comprehend informed consent
* Unwilling to sign informed consent
* Cognitive impairment, psychotic disorder or severe chronic mental health condition based on clinical intake DSM-V assessment
* Older than 65 years of age
* Reported suicidality in last 30 days
* Current prisoner
* Pregnant in the 3rd trimester
* Pregnant (MRI subsample only)
* Not willing to be audio recorded
* Not willing to have data stored for research purposes

Additional exclusion criteria for brain imaging sub-study:

* Older than 50 years of age
* Not in good general health
* Left handed (with a mean item score >1 on the handedness scale)
* Currently pregnant
* Current medical devices (cardiac pacemaker, implanted cardiac defibrillator, carotid artery vascular clamp, neurostimulator, cochlear implant, metal fragments (including shrapnel) in the head, eyes, or skin, vascular stent, ocular implant, penile implant, vascular filter for clots (including Greenfield, Umbrella, or Birds Nest filters)
* Other non-removable devices (IUD, dental braces or retainer, piercings that cannot be removed prior to resting, permanent eye-liner)
* Body Mass Index (BMI) greater than 36
* History of head trauma resulting in loss of consciousness for more than 5 minutes
* Documented or subjectively reported claustrophobia
* Having hair extensions or a wig connected by wire

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Black, PhD, MPH, Principal Investigator — University of Southern California
Locations (1):
- Prototypes' Pomona Women's Center, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Not until 12 months after final outcomes manuscript is submitted for publication. Contact davidbla@usc.edu for dataset
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data available from 2021 and for 5 years after contacting davidbla@usc.edu for shared files.
Access Criteria: Contact davidbla@usc.edu

REFERENCES:
- [Background] Amaro H, Spear S, Vallejo Z, Conron K, Black DS. Feasibility, acceptability, and preliminary outcomes of a mindfulness-based relapse prevention intervention for culturally-diverse, low-income women in substance use disorder treatment. Subst Use Misuse. 2014 Apr;49(5):547-59. doi: 10.3109/10826084.2013.852587. PMID 24611850
- [Background] Black DS, O'Reilly GA, Olmstead R, Breen EC, Irwin MR. Mindfulness-based intervention for prodromal sleep disturbances in older adults: design and methodology of a randomized controlled trial. Contemp Clin Trials. 2014 Sep;39(1):22-7. doi: 10.1016/j.cct.2014.06.013. Epub 2014 Jul 1. PMID 24993561
- [Background] Hanley A, Garland EL, Black DS. Use of mindful reappraisal coping among meditation practitioners. J Clin Psychol. 2014 Mar;70(3):294-301. doi: 10.1002/jclp.22023. Epub 2013 Jul 1. PMID 23818289
- [Background] Li MJ, Black DS, Garland EL. The Applied Mindfulness Process Scale (AMPS): A process measure for evaluating mindfulness-based interventions. Pers Individ Dif. 2016 Apr 1;93:6-15. doi: 10.1016/j.paid.2015.10.027. PMID 26858469
- [Background] Black DS, Slavich GM. Mindfulness meditation and the immune system: a systematic review of randomized controlled trials. Ann N Y Acad Sci. 2016 Jun;1373(1):13-24. doi: 10.1111/nyas.12998. Epub 2016 Jan 21. PMID 26799456
- [Background] Galla BM, O'Reilly GA, Kitil MJ, Smalley SL, Black DS. Community-Based Mindfulness Program for Disease Prevention and Health Promotion: Targeting Stress Reduction. Am J Health Promot. 2015 Sep-Oct;30(1):36-41. doi: 10.4278/ajhp.131107-QUAN-567. Epub 2014 Aug 27. PMID 25162319
- [Background] Garland EL, Black DS. Mindfulness for chronic pain and prescription opioid misuse: novel mechanisms and unresolved issues. Subst Use Misuse. 2014 Apr;49(5):608-11. doi: 10.3109/10826084.2014.852801. No abstract available. PMID 24611857
- [Background] Peltz L, Black DS. The thinking mind as addiction: mindfulness as antidote. Subst Use Misuse. 2014 Apr;49(5):605-7. doi: 10.3109/10826084.2014.852803. No abstract available. PMID 24611856
- [Background] Witkiewitz K, Black DS. Unresolved issues in the application of mindfulness-based interventions for substance use disorders. Subst Use Misuse. 2014 Apr;49(5):601-4. doi: 10.3109/10826084.2014.852797. No abstract available. PMID 24611855
- [Background] Black DS. Mindfulness-based interventions: an antidote to suffering in the context of substance use, misuse, and addiction. Subst Use Misuse. 2014 Apr;49(5):487-91. doi: 10.3109/10826084.2014.860749. PMID 24611846
- [Background] Black DS. Mindfulness and substance use intervention. Subst Use Misuse. 2012 Feb;47(3):199-201. doi: 10.3109/10826084.2011.635461. No abstract available. PMID 22217122
- [Background] Amaro H, Black DS. Mindfulness-Based Intervention Effects on Substance Use and Relapse Among Women in Residential Treatment: A Randomized Controlled Trial With 8.5-Month Follow-Up Period From the Moment-by-Moment in Women's Recovery Project. Psychosom Med. 2021 Jul-Aug 01;83(6):528-538. doi: 10.1097/PSY.0000000000000907. PMID 34213858
- [Result] Amaro H, Black DS. Moment-by-Moment in Women's Recovery: Randomized controlled trial protocol to test the efficacy of a mindfulness-based intervention on treatment retention and relapse prevention among women in residential treatment for substance use disorder. Contemp Clin Trials. 2017 Nov;62:146-152. doi: 10.1016/j.cct.2017.09.004. Epub 2017 Sep 14. PMID 28918120
- [Result] Black DS, Amaro H. Moment-by-Moment in Women's Recovery (MMWR): Mindfulness-based intervention effects on residential substance use disorder treatment retention in a randomized controlled trial. Behav Res Ther. 2019 Sep;120:103437. doi: 10.1016/j.brat.2019.103437. Epub 2019 Jul 7. PMID 31419610
- [Result] Kechter A, Amaro H, Black DS. Reporting of Treatment Fidelity in Mindfulness-Based Intervention Trials: A Review and New Tool using NIH Behavior Change Consortium Guidelines. Mindfulness (N Y). 2019 Feb;10(2):215-233. doi: 10.1007/s12671-018-0974-4. Epub 2018 Jun 22. PMID 30854147
- [Derived] Rivera D, Dueker D, Amaro H. Examination of referral source and retention among women in residential substance use disorder treatment: a prospective follow-up study. Subst Abuse Treat Prev Policy. 2021 Mar 2;16(1):21. doi: 10.1186/s13011-021-00357-y. PMID 33653374
- See also: American Mindfulness Research Association — https://goamra.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were adult women clinically diagnosed with SUD and admitted to residential SUD treatment. Recruitment spanned 2015-2018. All patients met one-on-one with the site's intake clinician coordinator. The site psychiatrist and on-site clinician coordinator discussed diagnostic assessment, determined final diagnoses, and made record in the patient chart. The site intake counselor verified study eligibility, and for those women who were eligible, informed clients about our study.
Pre-assignment Details: Of 367 potential participants who were screened for the study at the residential site, 200 were eligible and randomized to study conditions and attended the first treatment sessions. Those who missed the first study class session (class overview and introduction) were excluded from the study by design leaving N = 200 enrolled in the trial, 100 per condition.
Groups:
- Mindfulness Meditation [100 Enrolled]: Mindfulness-Based Relapse Prevention-Women (MBRP-W)
  Mindfulness Meditation: MBRP-W is delivered in 12 bi-weekly 80-minute group sessions. Facilitators with previous experience in MBSR and trained in MBRP-W will deliver each group. Each session has a central theme and is divided into five segments consisting of: (a) a welcome meditation or other mindfulness practice, (b) a review of session objectives, (c) a brief didactic psycho-educational presentation and discussion based on the session's theme, (d) experiential and formal meditation or other practices, and (e) readings and assignments for the next class. Participants are expected to learn skill building techniques to reducing stress using mindfulness-based principles to complement their recovery treatment program.
- Active Comparator [100 Enrolled]: Brain and Recovery (B&R)
  Brain and Recovery (B&R): B&R is delivered in 12 bi-weekly 80-minute group sessions delivered by two trained interventionists. The B&R group will receive didactic education on the neurobiology of addiction. B&R contains no information on behavior change, stress reduction, or mindfulness-based or relapse-related content. The intervention was developed over three years with a population similar to those in the study and with input from patients and experts on neurobiology of addiction. Topics include: (1) brain structures and functions related to addiction, (2) effects of various types of substances on the brain, and (3) rewarding effects and how these lead to addiction. Participants are expected to gain knowledge pertaining to the effects of drugs on the brain.
Period: Overall Study
Arm/Group | Mindfulness Meditation [100 Enrolled] | Active Comparator [100 Enrolled]
Started | 100 | 100
Completed | 87 | 93
Not Completed | 13 | 7
Not completed — Lost to Follow-up | 13 | 7

BASELINE CHARACTERISTICS:
Population: Women in SUD treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Meditation [100 Enrolled] | Active Comparator [100 Enrolled] | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (9.8) | 32.6 (8.4) | 32.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 60 | 116
  Not Hispanic or Latino | 43 | 38 | 81
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants] — Southern California
  participants
    United States | 100 | 100 | 200
SUD diagnosis DSM5 [Number; unit: participants] — Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition
  participants
    Alcohol use disorder | 10 | 9 | 19
    Drug use disorder | 71 | 74 | 145
    Both disorders | 18 | 14 | 32
    Missing | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Treatment Completion
Description: Number of women being designated by the site clinic as a completer during a discharge event.
Time Frame: 5 month follow period
Population: Women with SUD at a residential treatment site
Measure: Number; unit: Number of women
Arm/Group | Mindfulness Meditation | Active Comparator
Number analyzed (Participants) | 100 | 100
Number of women | 43 | 31
Statistical Analysis 1: Comparison: Mindfulness Meditation vs Active Comparator; 150 day period was selected for this outcome for a conceptual reason; that being, residential treatment average length of stay; Test type: Superiority; p < 0.05, Regression, Cox

2. Primary Outcome: Days of Any Drug Use
Description: Days of any drug use to include multiple drug types from study intervention end date to follow-up
Time Frame: 8.5 months
Population: Women with SUD enrolled in a residential treatment program who remained in the study and completed follow-up assessments approximately 8.5 months after the start of the intervention.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mindfulness Meditation | Active Comparator
Number analyzed (Participants) | 88 | 93
days | 16.92 (32.81) | 24.97 (51.65)
Statistical Analysis 1: Comparison: Mindfulness Meditation vs Active Comparator; Test type: Superiority; p < 0.05, Negative Binomial Hurdle Model

3. Secondary Outcome: Psychological Symptoms
Description: Five Facet Mindfulness Questionnaire (FFMQ): higher scores indicate better mindfulness qualities (better outcome).
  Perceived Stress Scale (PSS): higher scores indicate greater perceived stress (worse outcome).
  Depression Anxiety Stress Scale (DASS): higher scores indicate greater depression, anxiety, and stress (worse outcome).
  Distress Tolerance Scale (DTS): higher scores indicate greater distress tolerance (better outcome).
  Difficulties in Emotion Regulation Scale (DERS): higher scores indicate greater difficulties in emotion regulation (worse outcome).
  Penn Craving Scale (PCS): higher scores indicate greater craving (worse outcome).
  Positive and Negative Affect Schedule (PANAS) - Negative Affect subscale: higher scores indicate greater negative affect (worse outcome).
  Minimum and maximum values are not standardized.
Time Frame: 8.5 months
Population: Women with SUD
Measure: Mean (Standard Deviation); unit: score on a non-standardized scale
Arm/Group | Mindfulness Meditation | Active Comparator
Number analyzed (Participants) | 100 | 100
score on a non-standardized scale
  Five Facet Mindfulness Questionnaire (high better; range 5-195) | 83 (1.3) | 85 (1.2)
  Perceived Stress Scale (high worse; range 0-40) | 18 (0.7) | 17 (.06)
  Depression Anxiety Stress Scale (high worse; range 0-63) | 9 (.6) | 9 (.6)
  Distress Tolerance Scale (high better; range 1-5) | 3.3 (.1) | 3.2 (.1)
  Difficulties in emotion regulation scale (high worse, range 7-126) | 74 (2.4) | 74 (2.4)
  Penn Alcohol Craving Scale (high worse, range 1-7) | 1.6 (.2) | 1.4 (.2)
  Negative Affect Subscale (high worse, range 10-50) | 23 (.8) | 23 (.8)
Statistical Analysis 1: Comparison: Mindfulness Meditation vs Active Comparator; Test type: Superiority; p < 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: 8.5 months
Description: No serious adverse events to report from trial. The serious adverse events administration was managed by the PIs and by university IRB.
Groups:
- Mindfulness Meditation [100 Enrolled in Trial] Women Not Attending First Session Were Not Enrolled: Mindfulness-Based Relapse Prevention-Women (MBRP-W)
  Mindfulness Meditation: MBRP-W is delivered in 12 bi-weekly 80-minute group sessions. Facilitators with previous experience in MBSR and trained in MBRP-W will deliver each group. Each session has a central theme and is divided into five segments consisting of: (a) a welcome meditation or other mindfulness practice, (b) a review of session objectives, (c) a brief didactic psycho-educational presentation and discussion based on the session's theme, (d) experiential and formal meditation or other practices, and (e) readings and assignments for the next class. Participants are expected to learn skill building techniques to reducing stress using mindfulness-based principles to complement their recovery treatment program.
- Active Comparator [100 Enrolled in Trial] Women Not Attending First Session Were Not Enrolled: Brain and Recovery (B&R)
  Brain and Recovery (B&R): B&R is delivered in 12 bi-weekly 80-minute group sessions delivered by two trained interventionists. The B&R group will receive didactic education on the neurobiology of addiction. B&R contains no information on behavior change, stress reduction, or mindfulness-based or relapse-related content. The intervention was developed over three years with a population similar to those in the study and with input from patients and experts on neurobiology of addiction. Topics include: (1) brain structures and functions related to addiction, (2) effects of various types of substances on the brain, and (3) rewarding effects and how these lead to addiction. Participants are expected to gain knowledge pertaining to the effects of drugs on the brain.
Arm/Group | Mindfulness Meditation [100 Enrolled in Trial] Women Not Attending First Session Were Not Enrolled | Active Comparator [100 Enrolled in Trial] Women Not Attending First Session Were Not Enrolled
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT02977988/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT02977988/SAP_001.pdf
  • Informed Consent Form (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT02977988/ICF_002.pdf